CLINICAL TRIAL: NCT05235334
Title: Light House- Pilot Study Evaluating Mental Health Improvements After Using Home Phototherapy Device With UVB LEDs
Brief Title: Evaluating Mental Health Improvements After Using Home Phototherapy Device With UVB LEDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BeneSol, Inc. dba SOLIUS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: QR-TPL-042
Record Dates: First submitted 2022-01-17; First posted 2022-02-11 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-02

CONDITIONS: Usability; Quality of Life

STUDY DESIGN:
Intervention Model Description: All enrolled participants will use the SOLIUS home device.
Masking Description: No masking will be used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Device user (Experimental): Participant will engage in treatment with the MySOLIUS device, twice per week for 16 weeks
  Interventions: Device: MySOLIUS

INTERVENTIONS:
Device: MySOLIUS — MySOLIUS is a portable light therapy device that is designed to deliver a small amount of targeted ultraviolet B (UVB) light to trigger the body's natural production of vitamin D.

SUMMARY:
The primary objective of this study is to evaluate the satisfaction of users with the MySOLIUS device by a non-professional in a home use environment. The secondary objective of this study is to demonstrate the safety and effectiveness of the MySOLIUS device in the improvement of mood/quality of life score.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be screened to determine eligibility for study entry. Participants who meet the eligibility requirements will be sent a study device to use in their home environment. Prior to beginning treatment with the device, participants will fill out a quality of life questionnaire. Participants will use the device twice per week, once for treatment on the front side and once for treatment on the back side of the body. Participants will use the device twice a week for 16 weeks, for a total of 32 treatments. After the 16 week treatment duration, participants will fill out a final quality of life questionnaire and a device usability questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18 years or older with Fitzpatrick skin types 1,2,3,4,5 and 6.
* The patient can understand the information provided to them and who have given written informed consent to the study.
* The patient can understand and complete self-administered questionnaires.
* The patient is able and willing to follow study procedures.
* Women of child-bearing potential must confirm use of an effective contraceptive for 30 days prior to enrolling and continued use throughout the study or have a negative pregnancy test.

Exclusion Criteria:

* History of underlying photosensitivity.
* Subjects who are pregnant
* Patients that have granulomatous disorders (such as sarcoidosis).
* Use of medications that cause a photosensitivity reaction.
* History of skin cancer in the last 5 years.
* Patients with history of hypocalcemia (calcium <8.6mg%), hypercalcemia(calcium >10.6mg%).
* Taking drugs known to influence vitamin D metabolism, such as glucocorticoids,antiseizure medications, or HIV/AIDS medications.
* Patients with a history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease within 3 months.
* Intentional artificial UV exposure (e.g. tanning bed, UVB phototherapy use) in the last 60 days or planned use while participating in the study.
* Participation in an investigational drug study within 30 days of the screening.
* Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Satisfaction of Users with the device by a non-professional in a home use environment. | After study completion, 16 weeks
  Participants will be surveyed on their satisfaction with the MySOLIUS device on a scale of Strongly Disagree (1) to Strongly Agree (7)

SECONDARY OUTCOMES:
Increase in the quality of life scale. | Prior to starting treatment and after study completion, 16 weeks
  Participants will be surveyed on a variety of quality of life questions. Scores range from a minimum value of 0 to a maximum value of 1,300 with higher scores indicating a better quality of life.
Composite of adverse events and any skin changes | 16 weeks
  Participants will be asked weekly if they experience any adverse events or skin changes.

CONTACTS AND LOCATIONS:
Overall Officials: Jashin J Wu, MD, Principal Investigator — Office of Jashin Wu, M.D.; Chih-ho Hong, MD, Principal Investigator — Dr. Chih-ho Hong Medical Inc.
Locations (2):
- Office of Jashin J. Wu, MD, Irvine, California, United States
- Dr. Chih-ho Hong Medical Inc., Surrey, British Colimbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.